CLINICAL TRIAL: NCT06838871
Title: Effect of Inspiratory Muscle Training Combined With Abdominal Drawing-In Maneuver on Balance, Gait, and Pulmonary Function in Subacute Stroke Patients: A Randomized Controlled Trial
Brief Title: Effects of Inspiratory Muscle Training and Abdominal Drawing-In Maneuver on Balance, Gait and Pulmonary Function in Stroke Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Sahmyook University (Other)
Responsible Party: Principal Investigator, DOHYOUNG KIM, Physical Therapist, Sahmyook University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: SYU 2025-01-008
Record Dates: First submitted 2025-02-16; First posted 2025-02-21 (Actual); Last update posted 2025-12-26 (Actual); Status verified 2025-04

CONDITIONS: Subacute Stroke; Balance Deficits
Keywords: Inspiratory muscle training; balance; stroke; abdominal muscles; gait
MeSH Terms: conditions — Stroke

STUDY DESIGN:
Intervention Model Description: Prospective, parallel-group randomized study
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Inspiratory Muscle Training (IMT) with Abdominal Drawing-In Maneuver (ADIM) Group (Experimental): participants recieve in IMT using a threshold resistance device, starting at 30% of maximal inspiratory pressure and progressively increasing to 60% over four weeks. The ADIM is performed with verbal and manual guidance to ensure correct deep abdominal muscle engagement. Sessions are conducted five times per week for four weeks, with each session lasting 40 minutes (20 minutes for each intervention).
  Interventions: Behavioral: Inspiratory Muscle Training (IMT) with Abdominal Drawing-In Maneuver (ADIM) training
- Sham Inspiratory Muscle Training(IMT) with Abdominal Drawing-In Maneuver(ADIM) Group (Sham Comparator): participants recieve simulated IMT with minimal resistance while performing the same ADIM as the experimental group. This design ensures that any effects observed can be attributed to inspiratory muscle training rather than ADIM. Sessions are conducted five times per week for four weeks, with each session lasting 40 minutes (20 minutes for each intervention).
  Interventions: Behavioral: Sham Inspiratory Muscle Training (IMT) with Abdominal Drawing-In Maneuver (ADIM) training

INTERVENTIONS:
Behavioral: Inspiratory Muscle Training (IMT) with Abdominal Drawing-In Maneuver (ADIM) training — ADIM aims to enhance trunk stability by selectively activating the transversus abdominis. Participants begin in a supine position and practice drawing in their abdomen toward the spine while maintaining a stable trunk and pelvis. A therapist provides verbal instructions and manual guidance to ensure proper muscle activation.
  IMT is performed using the Threshold RMT device (IMT, GH INNOTEK, Busan, South Korea). Participants wear a nose clip and start with 30% of Maximal Inspiratory Pressure (MIP), gradually increasing by 10% per week to reach 60% MIP by the final week. Each session consists of five sets of 10-15 repetitions, with a one-minute rest between sets.
  Arms: Inspiratory Muscle Training (IMT) with Abdominal Drawing-In Maneuver (ADIM) Group
Behavioral: Sham Inspiratory Muscle Training (IMT) with Abdominal Drawing-In Maneuver (ADIM) training — Sham IMT with ADIM training performs the same ADIM protocol as the IMT with ADIM training but undergoes IMT with minimal resistance (0 cmH₂O) to prevent actual muscle strengthening. This design ensures that the effects observed can be attributed to IMT rather than ADIM.
  Arms: Sham Inspiratory Muscle Training(IMT) with Abdominal Drawing-In Maneuver(ADIM) Group

SUMMARY:
This study examines how Inspiratory Muscle Training (IMT) combined with the Abdominal Drawing-In Maneuver (ADIM) affects balance, gait, and breathing in stroke patients. It aims to determine whether this combined intervention improves mobility and respiratory function more effectively than standard rehabilitation.

DETAILED DESCRIPTION:
This study investigates the effects of Inspiratory Muscle Training (IMT) and Abdominal Drawing-In Maneuver (ADIM) on stroke rehabilitation. IMT involves resistance-based breathing exercises to strengthen the inspiratory muscles and improve pulmonary function, while ADIM focuses on activating the deep abdominal muscles, particularly the transversus abdominis, to enhance trunk stability and postural control. Participants in the intervention group perform IMT using a threshold resistance device, starting at 30% of MIP and progressively increasing to 60% MIP over four weeks. ADIM exercises are conducted with verbal and manual guidance to ensure proper engagement of core muscles. Sessions are held five times per week for four weeks, with each session lasting 40 minutes (20 minutes for each intervention). The control group receives conventional rehabilitation without resistance-based inspiratory training.

The study utilizes TIS, BBS and TUG to assess balance, FGA to evaluate gait performance, and MIP and MEP to measure respiratory function. Assessments are conducted before and after the intervention to evaluate changes resulting from the treatment.

Eligible participants are individuals with subacute stroke (onset within 1-6 months), an MMSE-K score of 24 or higher, and the ability to walk at least 6 meters with or without an assistive device. Exclusion criteria include conditions prohibiting the Valsalva maneuver (e.g., glaucoma, aneurysm, pulmonary hypertension), acute respiratory infections, severe cognitive or language impairments, prior inspiratory muscle training within the past six months, unstable medical conditions, and neurological or musculoskeletal disorders affecting gait and balance.

This study aims to determine whether the combined application of IMT and ADIM enhances functional recovery, improves postural control, and promotes better respiratory health in stroke patients. The findings may contribute to the development of more effective rehabilitation strategies for improving quality of life in individuals recovering from stroke.

ELIGIBILITY:
Inclusion Criteria:

* Participants diagnosed with subacute stroke (1-6 months post-onset)
* Mini-Mental State Examination-Korean (MMSE-K) score of 24 or higher
* Ability to walk at least 6 meters, with or without an assistive device

Exclusion Criteria:

* Conditions prohibiting the Valsalva maneuver (e.g., glaucoma, aneurysm, pulmonary hypertension)
* Acute respiratory infections
* Severe language or cognitive impairments preventing communication
* Previous inspiratory muscle training within the last 6 months
* Unstable medical conditions (e.g., uncontrolled hypertension, diabetes)
* Neurological disorders affecting function and balance (e.g., Parkinson's disease, multiple sclerosis)
* Severe musculoskeletal impairments limiting functional mobility.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2025-03-24 (Actual); Primary Completion 2025-04-25 (Actual); Study Completion 2025-10-21 (Actual)

PRIMARY OUTCOMES:
Change in Trunk Control as Measured by the Trunk Impairment Scale (TIS) | change from Baseline to 4 weeks post intervention
  The TIS assesses trunk stability, coordination, and dynamic sitting balance in participants. It consists of three subscales: static sitting balance (score range: 0-7), dynamic sitting balance (score range: 0-10), and trunk coordination (score range: 0-6). The total score ranges from 0 to 23, with higher scores indicating better trunk control. The test is conducted with the participant seated on a firm, stable surface without back or arm support.
Change in Functional Mobility as Measured by the Timed Up and Go (TUG) Test | change from Baseline to 4 weeks post intervention
  TUG Test assesses functional mobility and fall risk. Participants start seated, stand up at a signal, walk 3 meters, turn around, walk back, and sit down. The test is timed in seconds, with lower times indicating better mobility. A time exceeding 14 seconds suggests an increased fall risk.
Change in Balance Ability as Measured by the Berg Balance Scale (BBS) | change from Baseline to 4 weeks post intervention
  BBS evaluates balance and fall risk through 14 items, covering sitting, standing, and positional changes. Each item is scored from 0 (unable) to 4 (normal performance), with a total possible score of 0 to 56. Scores below 44 indicate a high fall risk.

SECONDARY OUTCOMES:
Change in Gait Performance as Measured by the Functional Gait Assessment (FGA) | change from Baseline to 4 weeks post intervention
  FGA evaluates dynamic walking ability. It consists of 10 tasks, including walking with head turns, speed changes, and obstacle navigation. Each item is scored from 0 (severe impairment) to 3 (normal performance), with a total possible score of 0 to 30. A lower score indicates greater functional impairment.
Change in Respiratory Muscle Strength as Measured by Maximal Inspiratory Pressure (MIP) and Maximal Expiratory Pressure (MEP) | change from Baseline to 4 weeks post intervention
  MIP and MEP measure respiratory muscle strength using a manometer (Pony Fx, Cosmed, Italy). MIP reflects diaphragm and inspiratory muscle strength, while MEP measures expiratory muscle power. Participants are seated, wear a nose clip, and perform three attempts with the highest value recorded.

CONTACTS AND LOCATIONS:
Locations (1):
- Zenith Hospital, Seoul, Seoul, South Korea

IPD SHARING:
Plan to Share IPD: No